CLINICAL TRIAL: NCT06188819
Title: Rolled Pericardium Versus Cryopreserved Allograft to Treat Native or Prosthetic Aortic Infection
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Paul Sabatier of Toulouse (Other)
Collaborators: LUCAS BATISTELLA, MD (Unknown); Kheira hireche, MD (Unknown); Ludovic CANAUD, MD PhD (Unknown)
Responsible Party: Principal Investigator, Aurélien Hostalrich, Clinical Professor, University Paul Sabatier of Toulouse
Other Study IDs: Infected Aorta
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Aortic Infections and Inflammations
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cryopreserved arterial allograft: Aortic infection treated by cryopreserved arterial allograft
  Interventions: Procedure: Explantation of a previous aortic graft or endograft and reconstruction by arterial allograft or rolled pericardium
- Rolled pericardium patch: Aortic infection treated by Pericardium patch rolled
  Interventions: Procedure: Explantation of a previous aortic graft or endograft and reconstruction by arterial allograft or rolled pericardium

INTERVENTIONS:
Procedure: Explantation of a previous aortic graft or endograft and reconstruction by arterial allograft or rolled pericardium — In situ reconstruction with explantation of the infected graft or endograft and reconstruction by allograft or pericardium

SUMMARY:
While surgery with anatomic reconstruction of prosthetic aortic infections and native infectious aortitis has become established over time, the ideal substitute is not clearly defined. The cryopreserved arterial allograft (AAC) recognized as resistant to infections not only presents availability problems making its use complicated, particularly in emergencies, with a certain number of long-term aneurysmal developments. The tubulized pericardium patch (PP), available in all cases, seems to give promising results in recent literature. The investigators propose a comparative study of these two substitutes in this indication.

We carried out a two-center observational study including retrospectively from January 2010 to July 2023 all patients operated on for aortic prosthesis infection and native infectious aortitis with AAC reconstruction and prospectively PP patch reconstructions from July 2018 to July 2023. The diagnosis of infection was established according to the MAGIC criteria. The patients' preoperative comorbidities were collected to compare the groups. Postoperative morbidity and mortality was then compared. The medium-term evaluation consisted of comparing according to the Kaplan Meier method: postoperative mortality, permeability, reinfection rate, reoperation rate.

ELIGIBILITY:
Inclusion Criteria:

* All aortic intervention performed for native aortic infection reconstruction with patch or allograft
* All aortic intervention performed for infected graft reconstruction with patch or allograft

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients operated on for a native infection or an aortic prosthesis who had pericardium or allograft reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2010-01-02 (Actual); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Mortality | day 30 post operative
  Number of patients death during post operative stay
Reintervention | 30 days, 6 months, 12 months, 24 months
  Rate of reintervention during post operative stay
Post operative Major cardiovascular adverse events (MACE) | day 30 post operative
  Rate of nonfatal stroke, nonfatal myocardial infarction, and cardiovascular death

SECONDARY OUTCOMES:
Permeability | 30 days, 6 months, 12 months, 24 months
  Rate of reintervention for occlusion of the patch or the allograft
Reinfection | 30 days, 6 months, 12 months, 24 months
  Rate of reintervention for infection of the patch or the allograft